CLINICAL TRIAL: NCT00406757
Title: Clinical Evaluation of 506U78 in Japanese Patients With Relapsed or Refractory T-cell Acute Lymphoblastic Leukemia or T-cell Lymphoblastic Lymphoma.
Brief Title: Clinical Evaluation of Nelarabine (506U78)in Japanese Patients With Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGA105446
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Leukaemia, Lymphoblastic, Acute and Lymphoma, Lymphoblastic
Keywords: T-cell; T-ALL; T-LBL; 506U78; ara-G; ara-GTP; Lymphoma; Leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — nelarabine

ARMS (5):
- Pediatric Arm 1 (Active Comparator): Cycle 1: Nelarabine 400mg/m2 will be administered once daily from Day 1 to Day 5 followed by 16 days of off-dose.
  Cycle 2 and subsequent Cycles: Nelarabine 650mg2 will be administered once daily from Day 1 to Day 5 followed by 16 days of off-dose.
  Interventions: Drug: Nelarabine injection 400mg/m2
- Pediatric Arm 2 (Active Comparator): Cycle 1 and subsequent Cycles: Nelarabine 650mg/m2 will be administered once daily from Day 1 to Day 5 followed by 16 days of off-dose.
  Interventions: Drug: Nelarabine injection 650mg/m2
- Adult Arm 1 (Active Comparator): Cycle 1: Nelarabine 1000mg/m2 will be administered once daily on Days 1, 3 and 5 followed by 16 days of off-dose.
  Cycle 2 and subsequent Cycles: Nelarabine 1500mg/m2 will be administered once daily on Days 1, 3 and 5 followed by 16 days of off-dose.
  Interventions: Drug: Nelarabine injection 1000mg/m2
- Adult Arm 2 (Active Comparator): Cycle 1 and subsequent Cycles: Nelarabine 1500mg/m2 will be administered once daily on Days 1, 3 and 5 followed by 16 days of off-dose.
  Interventions: Drug: Nelarabine injection 1500mg/m2
- Pediatric Arm 3 (Active Comparator): Nelarabine 650mg/m2 will be administered once a day from Day 1 to Day 5.
  Interventions: Drug: Nelarabine injection 650mg/m2

INTERVENTIONS:
Drug: Nelarabine injection 400mg/m2 — Cycle 1: Nelarabine 400mg/m2 will be administered once a day from Day 1 to Day 5.
  Cycle 2 and subsequent Cycles: Nelarabine 650mg/m2 will be administered once daily from Day 1 to DAy 5.
  Arms: Pediatric Arm 1
Drug: Nelarabine injection 650mg/m2 — Nelarabine 650mg/m2 will be administered once a day from Day 1 to Day 5.
  Arms: Pediatric Arm 2; Pediatric Arm 3
Drug: Nelarabine injection 1000mg/m2 — Cycle 1: Nelarabine 1000mg/m2 will be administered once a day on Days 1, 3 and 5.
  Cycle 2 and subsequent Cycles: Nelarabine 1500mg/m2 will be administered once a day on Days 1, 3 and 5.
  Arms: Adult Arm 1
Drug: Nelarabine injection 1500mg/m2 — Nelarabine 1500mg/m2 will be administered once a day on Days 1, 3 and 5.
  Arms: Adult Arm 2

SUMMARY:
In Japan, patients with relapsed or refractory T-ALL/T-LBL represent an extremely small patient population. While the small number of patients presents a practical limitation to the size of a clinical trial, patients whose disease has not responded to or has relapsed after treatment with multiple prior chemotherapy regimens have no accepted standard therapies available. Japanese leukemia experts have expressed interest in evaluating 506U78 in Japanese patients with relapsed or refractory T-ALL/T-LBL. In order to obtain safety, tolerability, and pharmacokinetic data of 506U78 in Japanese patients, this study is designed to maximize the contribution of each available patient.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytogenetic documented diagnosis of T-ALL or T-LBL.
* Disease that is refractory to at least one prior chemotherapy regimen, or has relapsed following complete remission to at least one prior chemotherapy regimen.
* At least 4 weeks since the last dose of prior last chemotherapy, or radiotherapy before beginning treatment with 506U78 (2 weeks is permitted if growth of blast cells is significant).
* Adequate function of other organ systems as measured as follows.Serum creatinine is less than 1.5 times of upper limit of normal and estimated creatinine clearance >=50 mL/min. Hepatic transaminases (SGPT and SGOT) <=3 x upper limit of normal, bilirubin is less than 1.5 times of upper limit of normal(<=5 x upper limit of normal if it is related by T-ALL or T-LBL).
* Adequate performance status (ECOG-PS<=2).
* Capable of giving informed consent which includes compliance with the requirements and restrictions listed in the consent form.
* Patient is willing to accept hospitalization during the blood sampling for pharmacokinetic measurement (i.e., Cohort 1: for pharmacokinetic sample collection during both cycle 1 and 2; and Cohort 2: for pharmacokinetic sample collection during cycle 1).
* Female subjects who are of child-bearing potential must have a negative pregnancy test at the Screening Visit and agree to utilize contraceptive methods during participation in the study and for at least six months following the last dose of 506U78 Injection. Female subjects may be defined as of non-child-bearing potential if they are physiologically incapable of becoming pregnant, including any female who is post-menopausal. For purposes of this study, postmenopausal is defined as one year without menses.

Exclusion Criteria:

* Active infection at time of treatment.
* Concurrent disease or condition that would make the subject inappropriate for study participation.
* Receiving any other anticancer agents or enrolled on any investigational study during the course of the study.
* Patients must have recovered to Grade I or less toxicity of all previous chemotherapy prior to treatment.
* History of seizure disorder within one year prior to the date of informed consent.
* Pregnancy (as demonstrated by a positive pregnancy test at pre-study/screening) or breastfeeding. Fertile women and men must practice adequate contraception throughout the study and at least 6 month after the last dose of study drug.

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08-30 (Actual); Primary Completion 2009-07-15 (Actual); Study Completion 2009-07-15 (Actual)

PRIMARY OUTCOMES:
Adverse events, changes from baseline in physical examination and clinical laboratory parameters12-lead ECGAssessment of pharmacokinetic endpoints of 506U78, ara-G and intracellular ara-GTP concentration. | Day 21

SECONDARY OUTCOMES:
Evaluation of response (e.g., CR, CR*) in patients with bone marrow involvement. | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Background] Horibe K, Takimoto T, Yokozawa T, Makimoto A, Kobayashi Y, Ogawa C, Ohno R, Koh N, Katsura K, Tobinai K. Phase I study of nelarabine in patients with relapsed or refractory T-ALL/T-LBL. Rinsho Ketsueki. 2011 Jun;52(6):406-15. PMID 21737993
- See also: Results for study 105446 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/PGA105446?search=study&search_terms=105446#rs